CLINICAL TRIAL: NCT02450708
Title: Selection of Allogeneic Hematopoietic Cell Donors Based on KIR and HLA Genotypes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Center for International Blood and Marrow Transplant Research (Network); Hackensack Meridian Health (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); M.D. Anderson Cancer Center (Other); Dana-Farber Cancer Institute (Other); University of Washington (Other); Mayo Clinic (Other); Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15-059
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Leukemia
Keywords: Allogeneic Hematopoietic Cell Donors; KIR and HLA Genotypes; 15-059
MeSH Terms: conditions — Leukemia

ARMS (2):
- For patients with 1 HLA-compatible donor for URD HCT (Experimental): For patients with 1 URD: donor KIR genotyping will be performed on the donor. Because donor selection will not depend on KIR/HLA genotyping, completion of donor KIR genotyping is not required prior to transplant.
  Interventions: Genetic: HLA genotyping
- For patients with >1 HLA-compatible donor for URD HCT (Experimental): For patients with 1 or more donor candidates, KIR genotyping may be performed for up to 5 donors. For patients with HLA-B alleles harboring the Bw4 epitope, KIR3DL1 allele typing will be performed at MSKCC.
  Interventions: Genetic: KIR genotyping; Genetic: HLA genotyping

INTERVENTIONS:
Genetic: KIR genotyping
  Arms: For patients with >1 HLA-compatible donor for URD HCT
Genetic: HLA genotyping

SUMMARY:
This study tests whether adding certain genetic factors to the process of picking a stem cell donor can decrease the chances that the patient's leukemia will come back after bone marrow transplantation. Stem cell donors are "matched" based on genes called human leukocyte antigens (HLA).

Currently, donors are selected largely on the basis of HLA gene typing alone. There is published data to show that donors with specific other genes called killer immunoglobulin-like receptors (KIR) may protect AML patients from having their leukemia return after a transplant. In this study, the best HLA matched donors will be tested for the KIR genes. If there is more than 1 donor available, a recommendation will be provided to study doctors as to which donors have potentially favorable KIR genes. The study doctors may or may not choose to use this donor for transplant or not based on his/her own judgment. Transplant care will not change otherwise as a result of this study.

This study is being done to demonstrate that AML patients who have donors with specific KIR and HLA genes will have a better outcome following transplant.

ELIGIBILITY:
Inclusion Criteria:

RECIPIENT

* Persons of all ages are eligible for this study.
* Patient must have diagnosis of acute myelogenous leukemia (AML) at MSK or a collaborating treating institution. Patients with de novo AML or AML with preceding myelodysplastic syndrome (MDS) are eligible.
* Patient must be a potential candidate for an unrelated transplantation procedure at the time of enrollment even though patient may not be eligible for transplantation in the future due to relapse or presence of co-morbidity(ies).
* An unrelated donor does not need to be identified at the time of enrollment. If an HLA-compatible unrelated donor is not identified for the patient, the patient will be removed from the study.

Exclusion Criteria:

* Recipients with an available sibling donor matched at HLA-A, HLA-C, and HLA-DRB1 (excluding identical twin siblings).
* Patients for whom post-transplant treatment is planned are not excluded from enrollment.
* Patients with prior allogeneic hematopoietic cell transplantation for AML. Note: Patients who have undergone prior hematopoietic cell transplantation for a diagnosis other than AML are still eligible for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
relapse | 1 year
  Demonstration of evidence of leukemia (>5% blasts in the bone marrow, peripheral blood blasts, or development of extramedullary disease) after initial achievement of either a CR or CRi.

SECONDARY OUTCOMES:
overall survival | 1 year
  Overall survival (OS). The time from study enrollment until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Hsu, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Moffitt Cancer Center, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Baylor University Medical Center, Dallas, Texas
  - Md Anderson Cancer Center, Houston, Texas
  - University of Washington School of Medicine, Seattle, Washington

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/